CLINICAL TRIAL: NCT06476457
Title: Low Cost, Low Intensity, Mobile-based Trauma Intervention (Facilitated STAIR Coach) for Use in Kenya
Brief Title: Use of Facilitated STAIR Coach in Kenya
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Kristina Korte, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024HSPH
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Facilatated STAIR Coach
Keywords: STAIR; STAIR Coach; post-traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: We will recruit 10 participants to assess the feasibility of using STAIR Coach mobile based app for PTSD in Kenya
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Facilitated STAIR Coach (Experimental): STAIR (Skills Training in Affective and Interpersonal Regulation ) Coach is a brief, low-intensity mobile-based intervention targeting difficulties in affective and interpersonal regulation. STAIR Coach participants will complete 10 interventions modules. Every two week, the participant will meet with a facilitator to review the module materials.
  Interventions: Behavioral: STAIR Coach

INTERVENTIONS:
Behavioral: STAIR Coach — STAIR is a brief, low-intensity intervention targeting difficulties in affective and interpersonal regulation that tend to be a significant problem for those exposed to traumatic events.
  Other Names: STAIR; Skills Training in Affective and Interpersonal Regulation

SUMMARY:
The specific aim of this project is to examine the feasibility of using a low cost, low intensity, mobile app-based intervention teaching emotion regulation and interpersonal skills to improve general well-being for those with probable post-traumatic stress disorder (PTSD) in Kenyan clinics.

DETAILED DESCRIPTION:
The aim of the present study is to examine the feasibility of the use of the Skills Training in Affective and Interpersonal Regulation (STAIR; Cloitre et al., 2020) Coach mobile app delivered through a mobile app for individuals with probable post-traumatic stress disorder (PTSD) in Kenya. This pilot study will recruit a total of 10 participants with probable PTSD. Participants will complete 10 modules focused on learning skills to improve interpersonal functioning and emotion regulation. The sessions will be facilitated by a mental health worker trained in STAIR. Participants will complete baseline (week 0), mid-treatmnet (week 5), post-treatment (week 11), one-month (week 15) and 3-month (week 23) follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* criteria

  1. 18 years of age or older
  2. ability to complete the study in English
  3. agreed to be contacted for follow-up studies when consenting to the parent study
  4. not currently enrolled in another form of psychotherapy
  5. if currently prescribed medications, participants must be on a stable dosage of psychotropic medications (i.e., prescribed on stable dose for 1 month or more)
  6. have a score of 33 or higher on the PCL-5 lifetime score in the parent study

     Exclusion Criteria:

  <!-- -->

  1. less than 18 years of age
  2. unable to complete the study in English
  3. did not agree to be contacted for follow-up studies when consenting to the parent study
  4. diagnosed with a psychotic disorder, unmedicated bipolar disorder, or severe substance-use disorder
  5. experiencing ongoing long-term trauma as it is a contraindication for trauma focused treatment
  6. experiencing acute levels of alcohol or is under the influence of an illegal substance, demonstrated by inpatient medical care for alcohol or substance abuse
  7. participant is not competent to consent to the study as measured by the UBACC in the parent study
  8. During parent study assessment (IRB23-0211), the participant receives a PCL score less than 33
  9. Participant is receiving inpatient psychiatric care at the time of the study or experiencing involuntary detention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for the DSM-5 (PCL-5) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  The PCL is an 18-item measure assessing symptions of post-trauamatic stress disorder. Higher scores indicate higher levels of trauma related symptoms.
Patient Health Questionnaire (PHQ-9) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  The PHQ-9 is a 9-item measure assessing symptoms of depression. Higher scores indicate greater levels of depressive symptoms.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  The PHQ-9 is a 9-item measure assessing symptoms of depression. Higher scores indicate greater levels of depressive symptoms.

IPD SHARING:
Plan to Share IPD: Undecided